CLINICAL TRIAL: NCT03309969
Title: Comparison of Intravascular Ultrasound With Venography in the Diagnosis and Treatment of Iliac Vein Compression Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2017-115
Record Dates: First submitted 2017-09-19; First posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-09

CONDITIONS: Iliac Vein Compression Syndrome
MeSH Terms: conditions — May-Thurner Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observation group: Subjects with suspicious iliac vein compression syndrome were included in the observation group.

SUMMARY:
The aim of this study is to compare intravascular ultrasound with venography in the diagnosis and treatment of iliac vein compression syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 90 years
* Willing to participate in and sign the informed consent
* Patients with suspicious iliac vein stenosis or compression presented by preoperative magnetic resonance venography (MRV)
* Patent common femoral vein and/or femoral vein of the study leg
* Undergoing iliofemoral venography with the intend to treat potential iliac vein compression syndrome

Exclusion Criteria:

* Not providing informed consent
* Venous compression caused by pelvic tumors or fibroid uterus
* Previous stent implantation or venovenous bypass surgery of the study leg
* Known metal allergy precluding the possibility of stent implantation
* Known iodine allergy or severe renal insufficient function which are unsuitable for venography
* Pregnant or planning to be pregnant recently
* Acute deep vein thrombosis or tumor thrombus involving the study leg
* Know history of thrombophilia (e.g. protein C or S deficiency, anti-thrombin III deficiency, etc )
* Any concurrent disease, for example, heart failure, might make the patients unsuitable for surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with suspicious iliac vein compression syndrome
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-10-30 (Estimated); Primary Completion 2018-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage diameter reduction | 1 month
  Compare the percentage diameter reduction measured by intravascular ultrasound (IVUS) and venography
Percentage area reduction | 1 month
  Compare the percentage area reduction measured by IVUS and the calculated percentage area reduction measured by venography

SECONDARY OUTCOMES:
CEAP score | 18 months
  Improvement in Clinical, Etiology, Anatomy, Pathophysiology (CEAP) score
Primary patency | 18 months
  Primary patency can be defined as without additional revascularization of the target lesions, the target vessels are still patent which measured by ultrasound or magentic resonance venography (MRV) and the diameter reduction is <50% during follow-up period.
Secondary patency | 18 months
  Secondary patency can be defined as: with additional revascularization of the target lesions after the first surgery in our department, the target vessels are still patent which measured by ultrasound or magentic resonance venography (MRV) and the diameter reduction is <50% during follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China